CLINICAL TRIAL: NCT04592783
Title: Postpartum Hypertension, Tight vs Liberal Control: A Randomized Controlled Trial
Brief Title: Postpartum Hypertension, Tight vs Liberal Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Oluyemi Aderibigbe, MD, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20200183
Record Dates: First submitted 2020-10-14; First posted 2020-10-19 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Hypertension in the Obstetric Context
Keywords: Postpartum; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Antihypertensive Agents

STUDY DESIGN:
Intervention Model Description: Multi-center Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight Blood Pressure Control (Experimental): Antihypertensive medications will be initialed once BP is at or above 140/90 mmHg
  Interventions: Drug: Antihypertensive Agents
- Liberal Blood Pressure Control (Experimental): Antihypertensive medications will be initialed once BP is at or above 150/95 mmHg
  Interventions: Drug: Antihypertensive Agents

INTERVENTIONS:
Drug: Antihypertensive Agents — Antihypertensive medications will be initialed once BP is at predetermined threshold

SUMMARY:
To determine if treatment of less severe hypertension in the postpartum period results in a lower frequency of maternal morbidity.

DETAILED DESCRIPTION:
Patients with postpartum hypertension are at risk of developing preeclampsia, eclampsia, and severe maternal morbidity. About one-third of eclampsia occurs in the postpartum period. Fifty percent of intra-cerebral hemorrhages occurring in association with preeclampsia occur in the postpartum period. In addition to the maternal morbidity that may arise from severe hypertension in the postpartum period, additional consequences of inadequate blood pressure control include maternal readmission, its associated costs to the healthcare system, and its destabilizing effect on a new family. Furthermore, pregnant women with hypertensive disorders in pregnancy are at an increased risk of persistent postpartum hypertension and metabolic syndrome within the first year after delivery. Therefore, untreated postpartum hypertension may significantly impact on long term cardiometabolic outcomes for reproductive aged-women.

Evidence-based guidance is lacking on the blood pressure threshold to initiate antihypertensive therapy in the postpartum period. Current clinical practice is extrapolated from management during pregnancy and no prior trials have been conducted on the threshold for initiation of antihypertensive medication in the postpartum period. A systematic review in 2017 concluded "there is a lack of good quality evidence for postpartum management, emphasizing the need for further RCTs directly comparing different antihypertensive agents, BP threshold for medication adjustment and different models of care, with outcome measures other than postnatal readmissions" Based on low quality evidence/expert opinion ACOG and the National Institute of Heath and Care Excellence (NICE) in the UK both recommend initiating antihypertensive at a BP threshold of 150/100mmhg. NICE further recommends keeping BP lower than 140/90mmHg in patients with chronic hypertension and reducing antihypertensive medications when BP is less than 130/80mmHg in this population. ACOG does not mention at which BP threshold to reduce medications or when to stop antihypertensive therapy. There are obvious gaps in knowledge as stated in the systematic review. Therefore, our objective is to provide evidence to inform best practices with regards to the management of hypertension in the postpartum period through this randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women aged 18-55 during delivery hospitalization.
* Diagnosis of gestational hypertension, preeclampsia without severe features, or chronic hypertension without requiring antihypertensive therapy who have Blood Pressure at/above 140/90 mmHg on 2 or more occasions more than 4 hours apart and do NOT meet criteria for preeclampsia with severe features and have not received any antihypertensive therapy during their hospitalization

Exclusion Criteria:

* History of chronic hypertension requiring antihypertensive therapy prior to or during pregnancy.
* Diagnosis and/or treatment of preeclampsia with severe features before trial enrollment
* Postpartum patients enrolled in another antihypertensive study (e.g CHAPS)
* Medical comorbidities including: Active connective tissue disease, chronic renal insufficiency, known cardiac disease or cerebrovascular disease.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 256 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
A composite of the following: Development of severe HTN or preeclampsia with severe features, hospitalization > 4 days, use of a second antihypertensive agent, adverse maternal outcomes and emergent treatment of severe HTN. | Within 2 weeks of hospital discharge
  Composite outcomes

SECONDARY OUTCOMES:
Hospital readmission secondary to HTN or preeclampsia in the first 14 days postpartum | 2 weeks
  Readmission
Persistence of hypertension (CHTN) at/beyond 14 days postpartum | 2 weeks
  Persistence of HTN
Medication side effects (hypotension | 2 weeks
  Side effects
Time to blood pressure control between different antihypertensive therapies | 2 weeks
  Time to BP control

CONTACTS AND LOCATIONS:
Overall Officials: Oluyemi Aderibigbe, MD, Principal Investigator — UH, Cleveland Medical Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Metrohealth Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No